CLINICAL TRIAL: NCT01499693
Title: Phase IIIb, Randomized, Triple-blinded and Crossover Study to Evaluate the Effect of Magnesium Pantoprazole 20mg Bid Versus Magnesium Pantoprazole 40mg qd on Intragastric Acid Inhibition Assessed by pHmetry, in Healthy Volunteers
Brief Title: Magnesium Pantoprazole 20mg b.i.d. vs Magnesium Pantoprazole 40mg q.d. on Intragastric Acid Inhibition
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MX026; U1111-1132-3320 (Registry Identifier: WHO)
Record Dates: First submitted 2011-09-12; First posted 2011-12-26 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Gastric pH Control
Keywords: Proton Pump Inhibitors; gastric pH

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnesium Pantoprazole 20mg (Experimental)
  Interventions: Drug: Magnesium Pantoprazole 20 mg
- Magnesium Pantoprazole 40mg (Active Comparator)
  Interventions: Drug: Magnesium Pantoprazole 40 mg; Drug: Placebo

INTERVENTIONS:
Drug: Magnesium Pantoprazole 20 mg — oral dose, twice a day
  Other Names: Tecta 20
  Arms: Magnesium Pantoprazole 20mg
Drug: Magnesium Pantoprazole 40 mg — oral dose, once a day (morning)
  Other Names: Tecta 40
  Arms: Magnesium Pantoprazole 40mg
Drug: Placebo — oral dose, once a day (night)
  Placebo will be administered at night in the group with 40mg magnesium pantoprazole to keep the blinding (so treatment administration is comparable w/the 20mg group).
  Arms: Magnesium Pantoprazole 40mg

SUMMARY:
The purpose of this study is to determine if magnesium pantoprazole 20 mg twice a day (b.i.d.), maintains gastric pH above 4 during a longer percentage of time than magnesium pantoprazole 40 mg once a day (qd). This is a comparison between split dose concept and standard dose of proton pump inhibitors.

DETAILED DESCRIPTION:
Eligible healthy volunteers will be randomly assigned for 2 different treatment sequences: A) magnesium pantoprazole 20 mg b.i.d. followed by magnesium pantoprazole 40 mg q.d. or B) magnesium pantoprazole 40 mg q.d. followed by magnesium pantoprazole 20 mg b.i.d.

Treatment sequences will be administrated as follows: 6 days with the first medication, followed by a washout period of 8 days (no medication) and a further period of 6 days with the second medication.

Treatment efficacy will be established by the percentage of time with intragastric pH >4, measured by 24-hour pH-Metry on day 6 of each medication (on-treatment measurement). Basal pH will be measured as reference.

The blinding distribution of treatments will be maintained for the patients, the doctor and the statistician who will analyze the data.

ELIGIBILITY:
Main inclusion criteria:

* Carlsson-Dent Questionnaire with score ≤ 4 (negative for GERD).
* Endoscopy: negative for GERD
* BMI between 18.5 and 30

Main exclusion criteria:

* Volunteers with any the following symptoms: dysphagia, digestive track bleeding, anorexia, anemia, involuntary weight loss.
* Women under breastfeeding period, pregnant or under pregnancy suspicion.
* Subjects with abnormal manometry (any motor esophageal disorder).
* Peptic ulcer history and/or ulcer complication.
* Volunteers under PPI treatment, H. pylori eradication treatment, H2 receptor antagonists, prokinetics or similar medication (current, during the last 30 days or during the trial).
* History of systemic glucocorticoids or non-steroidal anti-inflammatory drugs (NSAID) use, during the last 30 days.
* Abnormal laboratory parameters or vital signs, considered clinically relevant by the researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Change in Percentage of time with intragastric pH above 4.0, measured by continuous 24 hour intragastric pH-Metry. | Three 24-hour measurements will be performed: on day 0 (baseline) and on day 6 of each treatment period.
  Electrode will be placed in the gastric lumen, 10 cm below the lower esophageal sphincter. The percentage of time with pH >4.0 between both treatments will be compared.

SECONDARY OUTCOMES:
Vital signs, physical exploration and common laboratory tests (if required). | Day 0 (baseline) and day 6 of each treatment period.
  Safety will be established by monitoring these clinical criteria

CONTACTS AND LOCATIONS:
Overall Officials: Edgardo Suarez, MD, MSc, Principal Investigator — Clinic at Hospital Español de Mexico; Jose A Vargas, MD, MSc, Study Director — Takeda
Locations (1):
- Hospital Español de Mexico, Mexico City, Mexico City, Mexico